CLINICAL TRIAL: NCT06901518
Title: A Pilot, Open-Label Study to Assess the Effect of Galcanezumab-gnlm in Reducing the Frequency and Severity of Post-Traumatic, Migrainous Headaches
Brief Title: The Effect of Galcanezumab-gnlm on Post-Traumatic, Migrainous Headaches
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Charles Argoff, MD, Albany Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5843
Record Dates: First submitted 2025-03-27; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Post-Traumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache | interventions — erenumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Active treatment arm (Experimental): All participants are in the active treatment arm, which consists of subcutaneous injections of galcanezumab-gnlm. The first dose is the FDA-approved loading dose of 240mg (120mg injections into two separate subcutaneous sites). The second and third doses consist of a single 120mg subcutaneous injection of galcanezumab-gnlm.
  Interventions: Drug: Galcanezumab-Gnlm

INTERVENTIONS:
Drug: Galcanezumab-Gnlm — Subcutaneous injection
  Other Names: EMGALITY

SUMMARY:
The goal of this pilot, open-label clinical trial is to determine whether the addition of galcanezumab-gnlm to stable conventional headache treatment will reduce the number of monthly migraine days in participants who have experienced a traumatic brain injury and since developed post-traumatic, migrainous headaches. The main questions it aims to answer are:

* if galcanezumab-gnlm is effective in reducing the frequency and severity of post-traumatic headaches with migraine features in study participants
* if galcanezumab-gnlm reduces the impact of migraine on the daily life of the study participants

Participants will complete five clinic visits over the study. Study participants will

* complete a baseline visit including a HIT-6 Headache Impact Test score
* complete a headache diary for 4 weeks to record the frequency and severity of migrainous headaches and other information
* if determined to be eligible for the trial, undergo a brief physical exam and receive treatment with galcanezumab-gnlm, with a loading dose of 240mg delivered subcutaneously
* receive two subcutaneous treatments with galcanezumab-gnlm (120mg) 4 weeks apart
* complete a final study visit with a brief physical exam and HIT-6 Headache Impact Test score

DETAILED DESCRIPTION:
At study start, participants will review eligibility criteria with the investigator, undergo a physical exam, and review concomitant medications and medical history. Participants will be given a HIT-6 assessment as a baseline score. Participants will then be instructed to complete a headache diary over the next 4 weeks to record frequency and severity of migrainous headaches, changes to their health, and any other associated symptoms they have experienced. Participants will return for their second study visit at week four to review their headache diary results, ensure continued eligibility for the study based on their diary results, and undergo a brief physical exam. If participants are determined to be eligible, they will receive treatment with subcutaneous galcanezumab-gnlm in the clinic. Galcanezumab-gnlm 120mg and 240mg are FDA-approved for the treatment of chronic and episodic migraines. Participants will be observed following the treatment for 15 minutes to assess and record adverse reactions. They will also complete a HIT-6 score. The patient's vital signs will be rechecked following this 15 minute observation period. At the third study visit, week eight, participants will return to clinic to review their headache diary and any changes to their health or medications since the previous study visit. Participants will undergo a brief physical exam and a HIT-6 test and be injected with subcutaneous galcanezumab-gnlm and monitored for 15 minutes. This process will be repeated during the fourth study visit, week twelve, when participants receive their third and final subcutaneous injection of galcanezumab-gnlm. At the fifth and final study visit, week sixteen, a brief physical exam will be completed, headache diaries will be reviewed with the participant, and a final HIT-6 test will be administered, comparing this score to the previous HIT-6 scores.

Data will be collected throughout the study at the time of each visit, week 0 (study start), week 4, week 8, week 12, and week 16 (study end). During these visits, a HIT-6 score will be completed in clinic to determine the impact that post-traumatic, migrainous headaches have on participants' daily lives. Additionally, headache diaries will be completed by study participants between each visit, and these diaries will be reviewed by the investigator at each visit to further clarify the impact that galcanezumab-gnlm has on overall reduction in post-traumatic, migrainous headache frequency and severity. Headache diaries will reflect the new occurrence and increase or decrease in associated symptoms experienced throughout the twenty-eight -day period between each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Documented history of traumatic brain injury (TBI); acceptable TBI diagnoses could include concussion, SDH, ICH, and/or SAH diagnosed using ICD-10 coding by a medical professional.
2. Frequent post-traumatic headaches with migraine features as defined by the International Classification of Headache Disorders, 3rd Edition (ICHD-3), and this must be documented using ICD-10 coding by a medical professional.
3. Able to consent and participate in this research study.
4. 18 years of age or older.
5. Trial participants may also be using a stable dose of one migraine preventative medication recognized by AHS/AAN as level A or B, for at least 4 months prior to the start of the study screening and start date. Participants should remain on this stable dose throughout the study.
6. Participants who are being treated with OnabotulinumtoxinA and still meet criteria for migraine preventative treatment will be allowed to enroll.
7. Participants may have focal neurologic deficits as a result of suffering a TBI.
8. After review of the headache diary completed during the baseline period, the participant can be classified by the investigator as experiencing either chronic or episodic migraine; Chronic migraine is characterized by the participant having 15 or more headache days, at least 8 of which classify as a migraine. Episodic migraine is characterized by the participant having fewer than 15 headache days per month, and at least 4 of these headache days would classify as migraine.

Exclusion Criteria:

1. Under 18 years of age
2. Participant has a history of migraine headaches, diagnosed via ICD-10 coding and as defined by ICHD-3 criteria, occurring prior to the traumatic brain injury.
3. Participant is not experiencing headaches with migrainous features as defined by the ICHD-3 criteria.
4. Participant is pregnant or lactating or planning on becoming pregnant within the next six months.
5. Participant is unable to give consent to participate.
6. Participant began using unconventional interventions or devices aimed at reducing migraines, like nerve blocks and transcranial magnetic stimulation, within the 2 months prior to study screening.
7. Participant is using opioid or barbiturate therapies on 5 or more days during pre-intervention period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Mean change in number of migraine days per month | 16 weeks
  To determine the mean change in number of migraine days per month at study end compared to baseline pre-injection 4-week period

SECONDARY OUTCOMES:
Headache frequency and severity | 16 weeks
  Headache frequency and severity as reported in the headache diary
Mean change in headache days per month | 8 weeks and 12 weeks
  Mean change in headache days per month at 8 weeks and 12 weeks compared to baseline
Mean change in HIT-6 score | 16 weeks (study end)
  Mean change in Headache Impact Test (HIT-6) score from baseline
Mean change in average number of days that acute headache medications used per month | 8, 12, and 16 weeks
  Mean change in average number of days that acute headache medications were used per month as reported in the 8, 12, and 16 week appointment, compared to baseline data

CONTACTS AND LOCATIONS:
Overall Officials: Charles Argoff, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No